CLINICAL TRIAL: NCT05361291
Title: Comparative Evaluation of Adding Dexamethasone to 2% Lidocaine (With and Without Epinephrine) on the Anesthetic Success Rate of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Evaluation of the Effect of Adding Dexamethasone to 2% Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexamethasone
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Lidocaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inferior Alveolar nerve block with 2% lidocaine with 1:80 000 epinephrine (Active Comparator): An Inferior Alveolar nerve block was given with 2% lidocaine with 1:80 000 epinephrine
  Interventions: Drug: Lidocaine Hydrochloride
- Inferior Alveolar nerve block with 2% lidocaine with 1:80 000 epinephrine with 2mg dexamethasone (Experimental): An Inferior Alveolar nerve block was given with 2% lidocaine with 1:80 000 epinephrine mixed with 2mg dexamethasone
  Interventions: Drug: Lidocaine Hydrochloride
- Inferior Alveolar nerve block with plain 2% lidocaine mixed with 2mg dexamethasone (Experimental): An Inferior Alveolar nerve block was given with plain 2% lidocaine mixed with 2mg dexamethasone
  Interventions: Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Inferior alveolar nerve block
  Other Names: dexamethasone

SUMMARY:
This randomized, double-blind clinical trial aimed at the evaluation of the effect of adding dexamethasone to 2% lidocaine, given as inferior alveolar nerve block in the endodontic management of symptomatic irreversible pulpitis. One hundred and twenty four patients received one of the three IANB injections before the endodontic treatment: 2% lidocaine with 1:80 000 epinephrine; 2% lidocaine with 1:80 000 epinephrine mixed with 2mg dexamethasone; and plain 2% lidocaine mixed with 2mg dexamethasone. The anesthetia was considered successful if the patients experienced no pain or faint/weak/mild pain during root canal access preparation and instrumentation (HP VAS score <55 mm). The effect of intraligamentary injections on maximum heart rates was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* absence of any periapical radiolucency on radiographs, except for a widened periodontal ligament
* active pain in a mandibular molar
* prolonged response to cold testing with an ice stick and an electric pulp tester
* vital coronal pulp on access opening and ability to understand the use of pain scales

Exclusion Criteria:

* a history of known or suspected drug abuse
* history of active peptic ulcer within the preceding 12 months
* history of bleeding problems or anticoagulant use within the last month
* known allergy, sensitivity, or contraindications to any opioid or nonopioid analgesic including aspirin or NSAIDs
* patients who had taken NSAIDs within 12 h before administration of the study drugs
* patients who were pregnant or breast-feeding

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Anesthtic success | 15 minutes after the inferior alveolar nerve block
  Pain during the endodontic treatment was assessed using a visual analog scale (Heft-Parker VAS). Success was defined as no or mild pain (pain score≤54mm on Hp VAS) during access preparation and root canal instrumentation.

SECONDARY OUTCOMES:
Heart Rate | After 1 minutes of initial injection
  The effect of injections on maximum heart rates was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Jamia MIliia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately after publication
Access Criteria: Immediately after publication